CLINICAL TRIAL: NCT03079206
Title: Correlation of the in Vivo Food Provocation Test With the in Vitro Basophile Activation Test in Hazelnut Allergic Patients
Brief Title: Basophile Activation Testing (BAT) in Hazelnut Allergy (Hazelnut BAT Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ADR-AC Laboratory, Berne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-02152
Record Dates: First submitted 2017-02-20; First posted 2017-03-14 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Food Allergy
Keywords: hazelnut; allergens; basophile-activation-test; food; allergy
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity | interventions — Skin Tests; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The study intends to compare the outcome of food challenge with hazelnut and the in vitro basophile activation test using hazelnut extract and allergens
Masking Description: In terms of study inclusion there will be no masking. Only the food challenge itself will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hazelnut allergy (Experimental): patients with positive case history of hazelnut allergy and a positive skin testing are undergoing a food challenge and blood sampling for basophile activation testing
  Interventions: Diagnostic Test: Food challenge; Diagnostic Test: skin testing; Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: Food challenge — food challenge with hazelnut
Diagnostic Test: skin testing — Skin testing with hazelnut extract
Diagnostic Test: blood sampling — blood sampling to perform basophile activation tests

SUMMARY:
The proposed study intends to compare the outcome of food challenge in hazelnut allergic patients with the outcome of basophile activation tests using hazelnut extract and components.

DETAILED DESCRIPTION:
Accurate diagnosis of food allergy depends on food challenge outcome. The proposed study intends to compare the outcome of food challenge in hazelnut allergic patients with the outcome of basophile activation tests using hazelnut extract and components to evaluate the diagnostic utility of basophile activation testing.

With a view towards improved in vitro diagnostic methods, the investigators intend to evaluate the diagnostic potential of basophile activation testing in patients with hazelnut allergy confirmed by a positive provocation or supported by a convincing history of anaphylactic reaction(s) to hazelnut in the past, patients with pollinosis but no symptoms of hazelnut allergy and non-atopic control subjects.

ELIGIBILITY:
Inclusion Criteria:

Primary Inclusion criteria:

* Male and female subjects, age ≥ 14 years
* Informed Consent as documented by signature

Secondary inclusion criterion

* Group A: positive case history of allergic reaction(s) to hazelnut positive double-blind placebo-controlled food challenge with hazelnut or positive titrated open food challenge with hazelnut or unambiguous case history of an anaphylactic reaction after hazelnut will be included without provocation
* Group B:positive skin test (SPT) with birch pollen and hazelnut and negative food provocation with hazelnut.
* Group C: negative case history of hazelnut and birch allergy and negative skin test (SPT) with hazelnut and birch pollen and negative food provocation with hazelnut

Exclusion Criteria:

* Drugs not allowed due to interference with the food challenge (or shortest interval between last treatment and food challenge): corticosteroids systemically (2 weeks), antihistamines (3 days), beta blocker (1 day), angiotensin converting enzyme (ACE) inhibitors (2 days), omalizumab (2 months)
* Women who are pregnant
* Lack of safe contraception
* Uncontrolled asthma, forced expiratory volume (1 second) <70% predicted value
* Acute allergic disease
* Chronic urticaria
* Mastocytosis
* Other clinically significant concomitant disease states
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with challenge confirmed food allergy to hazelnut and a positive basophile activation test | up to 3 years
  outcome of food challenge in hazelnut allergic patients will be compared to the outcome of basophile activation using hazelnut extract and allergens

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ballmer-Weber, Prof., Principal Investigator — Allergy Unit, Department of Dermatology, University Zürich
Locations (1):
- Allergy Unit, Department of Dermatology, University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No